CLINICAL TRIAL: NCT00870259
Title: An Investigation of Physiological Adaptations Contributing to Weight Regain After Weight Loss
Brief Title: Investigating Physiological Adaptations to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Priya Sumithran, Clinical research fellow, University of Melbourne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP 508920
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Weight loss; Weight maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Optifast VLCD — Meal replacement, three times daily for 8 weeks

SUMMARY:
The purpose of this study is to examine the effect of diet-induced weight loss on the levels of circulating nutrients and hormones which are involved in feelings of hunger and satiety.

ELIGIBILITY:
Inclusion Criteria:

* males and post-menopausal females
* aged over 18 years
* BMI 27-40kg/m2
* weight-stable

Exclusion Criteria:

* major comorbid medial condition (including diabetes)
* taking medications known to affect weight
* smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Difference in fasting and/or post-prandial hormone levels following weight loss and after weight maintenance compared with baseline | 2, 6 and 12 months

SECONDARY OUTCOMES:
Difference in fasting and/or post-prandial hormone levels in ketotic compared with non-ketotic state | week 8 vs week 10
Correlation of fasting and post-prandial hormone levels with ratings of hunger and satiety | 0, 2, 6 and 12 months
Association of psychosocial factors with successful weight maintenance | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg Repatriation Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981